CLINICAL TRIAL: NCT06423183
Title: Interprofessional Mindfulness Practices Advancing Cancer Teamwork (IMPACT Study)
Brief Title: Interprofessional Mindfulness Practices Advancing Cancer Teamwork
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0517; A539713 (Other: UW Madison); Protocol Version 6/17/2024 (Other: UW Madison); UW24074 (Other: WISC OnCore)
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Burn Out
Keywords: oncology; health care; clinicians; mindfulness; well-being
MeSH Terms: conditions — Burnout, Psychological; Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a prospective, pre-post study at a single institution
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-Based Team Resilience Training (Experimental)
  Interventions: Behavioral: A Mindful Approach to Building a Resilient Healthcare Workforce (RENEW)

INTERVENTIONS:
Behavioral: A Mindful Approach to Building a Resilient Healthcare Workforce (RENEW) — Synchronous, 4-month intervention that teaches skills in mindfulness, stress management, and resilience as an individual and as a team. Sessions occur monthly and include a 1 hour in-person introductory session followed by 3 50-minute virtual sessions.

SUMMARY:
The purpose of the research is to understand if mindfulness team training can improve the well-being and teamwork in caring for oncology patients. This study will enroll healthcare professionals in oncology teams, including clinic nurses, nurse managers, medical assistants, social workers, technicians, patient navigators, advanced practice providers, and physicians at UW Madison. Participants will be on study for up to approximately 6 months.

DETAILED DESCRIPTION:
Aim 1: Determine the effect of resilience training on team resilience and well-being. The investigators test the hypothesis that resilience training provided to interprofessional oncology care teams will improve team resilience and individual well-being.

Aim 2: Determine the feasibility and acceptability of a resilience training on team resilience. The investigators test the hypothesis that resilience training is feasible and acceptable in interprofessional oncology care teams.

ELIGIBILITY:
Inclusion Criteria:

* A care provider in an oncology clinic team (clinic nurse, nurse manager, medical assistant, technician, social worker, patient navigator, advanced practice provider, physician)

Exclusion Criteria:

* Does not participate in patient care or support services

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-09-26 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Teamwork Measure | baseline (pre-intervention), post-intervention (3 months), follow up (6 months)
  4-item Edmondson's psychology safety scale is scored on a likert scale from 1 (strongly disagree) to 7 (strongly agree), where higher scores indicate higher psychology safety
Number of Participants Who Attend Each Session | up to 3 months
  Session 1 baseline, session 2 at 1 month, session 3 at 2 months, session 4 at 3 months
Acceptability of Intervention Measure (AIM) | up to 3 months
  AIM is a 4-item survey scored on a 5 point likert scale from 1 (completely disagree) to 5 (completely agree), where higher scores indicate greater acceptability.
Intervention Appropriateness Measure (IAM) | up to 3 months
  IAM is a 4-item survey scored on a 5 point likert scale from 1 (completely disagree) to 5 (completely agree), where higher scores indicate greater appropriateness.
Feasibility of Intervention Measure (FIM) | up to 3 months
  FIM is a 4-item survey scored on a 5 point likert scale from 1 (completely disagree) to 5 (completely agree), where higher scores indicate greater feasibility.

SECONDARY OUTCOMES:
Change in Stress measured by Perceived Stress Scale (PSS) | baseline (pre-intervention), post-intervention (3 months), follow up (6 months)
  PSS is a 10-item survey scored from 0 (never) to 4 (very often) for a total possible range of scores from 0-40 where higher scores indicate higher perceived stress.
Change in Burnout measured by Maslach Burnout Inventory | baseline (pre-intervention), post-intervention (3 months), follow up (6 months)
  This is a 2-item survey scored from 0-6 where higher scores indicate increased burnout.
Change in Resilience measured by Connor Davidson Resilience Scale (CD-RISC 2) | baseline (pre-intervention), post-intervention (3 months), follow up (6 months)
  CD-RISC 2 is a 2-item survey each scored on a 5 point likert scale from 0 (not true at all) to 4 (true nearly all of the time), higher scores indicate increased resilience.
Change in Well-being measured by Flourishing Index | baseline (pre-intervention), post-intervention (3 months), follow up (6 months)
  Flourishing measure is a 12-item survey that measure well being in each of 6 domains: happiness and life satisfaction; mental and physical health; meaning and purpose; character and virtue; close social relationships; financial and material stability. Each domain is scored from 0 - 10 where higher numbers are indicative of increased well being.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Wilke, MD, FACS, Principal Investigator — UW Carbone Cancer Center
Locations (1):
- UW Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT06423183/ICF_000.pdf